CLINICAL TRIAL: NCT02923219
Title: The Clinical Application of Adipose-Derived Stem Cells on Facial Rejuvenation
Acronym: ADSCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Peisheng, Vice-President of the Affiliated Hospital of Xuzhou Medical College, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL020-01
Record Dates: First submitted 2016-08-22; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Facies
Keywords: Facial Rejuvenation; Adipose-Derived Stem Cells
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cells separation (Experimental): Stem cells separation: The adipose-derived stem cells are separated from vacuumed fat obtained through liposuction of abdomen, hip, thigh and so on. It was confirmed the adipose-derived stem cells can be induced differentiation into fat cells under the special condition in the current literature.Stem cells are used to treat wrinkles and facial rejuvenation.
  Interventions: Biological: Adipose-derived stem cells

INTERVENTIONS:
Biological: Adipose-derived stem cells — The adipose-derived stem cells therapy involve injection of patient's own adipose-derived stem cells. Local anesthetic will be applied to the face prior to the injection. For adipose-derived stem cells preparation, proper volume of fat cells will be collected from each patient just before each procedure. The stem cells will be injected into each standardized injection point in a superficial manner. The injections points are along the inferior border of cheek and mid-cheek and temple, where will be followed by 10-15 minutes of icing.

SUMMARY:
The purpose of this study is to determine whether the adipose-derived stem cells therapy is effective in the treatment of facial rejuvenation.

DETAILED DESCRIPTION:
This study will be a prospective study of patients who undergo adipose-derived stem cells therapy for facial rejuvenation at the hospital of Xuzhou medical university. The therapy involves injection of patient's own adipose-derived stem cells, which are separated from vacuumed fat obtained through liposuction of abdomen, hip, thigh and so on. It was confirmed the adipose-derived stem cells can be induced differentiation into fat cells, osteoblasts, chondrocytes, muscle cells, endothelial cells and so on under the corresponding condition in the current literature. The therapy has evolved as a less invasive technique for facial rejuvenation compared to more traditional techniques，such as fat cells injection, sodium hyaluronate injection. Through the use of pre and post treatment photos, three-dimensional skin CT, in addition to the therapeutic evaluation, patient satisfaction questionnaire and a clinician assessment, it is our hope that the investigators will confirm the rejuvenating capabilities of adipose-derived stem cells therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages18-60
* Patients of all racial and ethnic origins
* Patients of all undergoing facial rejuvenation

Exclusion Criteria:

* Ages under 18, and above 60
* Female patients in pregnancy or menstrual period
* Patients undergoing facial rejuvenation using other methods including botox injections, chemical peels, face lifts and others
* Patients using blood thinners, aspirin and hormone, that cannot be stopped
* Patients suffering with severe organic disease, such as coronary heart disease, hypertension, diabetes, lung dysfunction and so on
* Patients suffering with mental disease, and acute or chronic infectious diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The therapeutic evaluation of adipose-derived stem cells or fat cells solely on facial rejuvenation | 1,3 and 6 Months Post-Surgery
  With the therapeutic evaluation of adipose-derived stem cells and fat cells solely on facial rejuvenation separately, which can reduce wrinkle and augment collagen of face skin. In order to assess the therapeutic effect, the investigators take face photos/make three-dimensional skin CT of face to evaluate the wrinkle and collagen before the therapy. Then take photos of face/ make three-dimensional skin CT of face to evaluate the wrinkle and collagen/ take patient satisfaction questionnaire and clinician assessment in 1 Months post-surgery. Take photos of face/ make three-dimensional skin CT of face/ take patient satisfaction questionnaire and clinician assessment in 3 Months post-surgery. Then take photos of face/ make three-dimensional skin CT of face to evaluate the wrinkle and collagen/ take patient satisfaction questionnaire and clinician assessment in 6 Months post-surgery. The investigators will summarize the therapeutic effect of facial rejuvenation based on the data.

SECONDARY OUTCOMES:
The therapeutic evaluation of adipose-derived stem cells combined with fat cells on facial rejuvenation | 1,3 and 6 Months Post-Surgery
  With the therapeutic evaluation of adipose-derived stem cells combined with fat cells on facial rejuvenation.The investigators take photos of face before the therapy and in 1, 3 and 6 Months Post-Surgery, take three-dimensional skin CT of face to evaluate the wrinkle and collagen and so on at the time points of pre-surgery and in 1, 3 and 6 Months post-surgery. In addition to the therapeutic evaluation, take patient satisfaction questionnaire and clinician assessment in 1, 3 and 6 Months post-surgery. The multiple measurements will be aggregated to arrive at facial rejuvenation. Compare the secondary outcome with primary outcome, then it can summarize the best method of facial rejuvenation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Peisheng, Principal Investigator — the Affiliated Hospital of the XuZhou Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hetherington HE, Block JE. Facial fat grafting with a prototype injection control device. Clin Cosmet Investig Dermatol. 2013 Sep 13;6:201-9. doi: 10.2147/CCID.S47469. eCollection 2013. PMID 24049453
- [Background] Winters R, Moulthrop T. Is autologous fat grafting superior to other fillers for facial rejuvenation? Laryngoscope. 2013 May;123(5):1068-9. doi: 10.1002/lary.23614. No abstract available. PMID 23619619
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Background] Yilgor Huri P, Cook CA, Hutton DL, Goh BC, Gimble JM, DiGirolamo DJ, Grayson WL. Biophysical cues enhance myogenesis of human adipose derived stem/stromal cells. Biochem Biophys Res Commun. 2013 Aug 16;438(1):180-5. doi: 10.1016/j.bbrc.2013.07.049. Epub 2013 Jul 20. PMID 23876311
- [Background] Shi Z, Neoh KG, Kang ET, Poh CK, Wang W. Enhanced endothelial differentiation of adipose-derived stem cells by substrate nanotopography. J Tissue Eng Regen Med. 2014 Jan;8(1):50-8. doi: 10.1002/term.1496. Epub 2012 May 24. PMID 22628362
- [Background] Salgado AJ, Reis RL, Sousa NJ, Gimble JM. Adipose tissue derived stem cells secretome: soluble factors and their roles in regenerative medicine. Curr Stem Cell Res Ther. 2010 Jun;5(2):103-10. doi: 10.2174/157488810791268564. PMID 19941460
- [Background] Li Q, Zhang A, Tao C, Li X, Jin P. The role of SDF-1-CXCR4/CXCR7 axis in biological behaviors of adipose tissue-derived mesenchymal stem cells in vitro. Biochem Biophys Res Commun. 2013 Nov 22;441(3):675-80. doi: 10.1016/j.bbrc.2013.10.071. Epub 2013 Oct 30. PMID 24184476
- [Derived] Yin Y, Li J, Li Q, Zhang A, Jin P. Autologous fat graft assisted by stromal vascular fraction improves facial skin quality: A randomized controlled trial. J Plast Reconstr Aesthet Surg. 2020 Jun;73(6):1166-1173. doi: 10.1016/j.bjps.2019.11.010. Epub 2019 Nov 29. PMID 32269011